CLINICAL TRIAL: NCT00232336
Title: Efficacy of Quetiapine in the Reduction of Cocaine Use and Cravings in Individuals With Cocaine Dependence
Brief Title: Quetiapine for Cocaine Use and Cravings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA 1 26; IRUS QUET0297
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine; drug; substance; abuse; addiction; dependence; quetiapine; antipsychotic; treatment
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Behavior, Addictive | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: quetiapine

SUMMARY:
The purpose of this study was to collect pilot data on whether quetiapine may be effective in the reduction of cocaine use and cravings in cocaine dependent individuals.

DETAILED DESCRIPTION:
Dopaminergic and serotonergic neurotransmitter systems are involved in cocaine use and cravings. Atypical antipsychotics act on these neurotransmitter systems, and therefore, may be beneficial in the treatment of cocaine addiction. This open label study assessed the efficacy of quetiapine for the treatment of cocaine use and craving in non-psychotic, cocaine dependent participants over 6 weeks of treatment. The primary outcome measures included self-report of cocaine use and self-report of cocaine cravings. This study also evaluated whether the severity of addiction predicts quetiapine efficacy.

Males and females, ages 18 - 65, with a DSM IV diagnosis of cocaine dependence were recruited for an open label trial of quetiapine dosed at 300-600 mg/day, with a target dose of 600 mg/day. Subjects were followed at weekly study visits to monitor general psychiatric and physical status, medication compliance, efficacy, and adverse events. Study participation included psychiatric and medical examinations, an electrocardiogram, an eye exam, laboratory tests, urine drug screens, electrocardiograms, and psychiatric and substance abuse interviews.

Twenty-three males were initiated on quetiapine treatment, the following results include the first twenty-two study completers. Twenty-two males (36-56 years) diagnosed with cocaine dependence without a psychotic disorder, were initiated on a six-week, open-label trial of quetiapine, 300-600 mg/day (QHS). Five participants discontinued prior to completing the first week of treatment, and 14 of 22 subjects completed the study. The mean dose of quetiapine was 429 mg/day. An intent-to-treat analysis found a significant decrease in cravings on the Brief Substance Craving Scale after six weeks (p < 0.01, Cohen's d = 1.23; repeated measures mixed effects random regression). Cocaine use, addiction severity, and psychopathology also decreased numerically, but not statistically, from baseline to end of study. Adverse effects were generally mild. Addiction severity did not predict quetiapine efficacy. Four subjects withdrew due to sedation; 2 were discontinued by the investigators, and 2 were lost to follow up. Study completers experienced a statistically significant mean weight gain of approximately 4.60 (95% CI, -6.05 - 3.17 kg)(mean baseline weight 86.9 (SD 18.38) kg).

Quetiapine treatment appears to have improved cocaine dependence, specifically cocaine cravings, in non-psychotic individuals. The observed weight change may reflect both weight gain associated with cocaine dependence and medication side effect. Controlled research is warranted to better define the potential role for quetiapine in the treatment of cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* DSM-IV diagnosis of cocaine dependence without psychotic symptoms
* Psychiatrically stable as evidenced by no psychiatric hospitalizations and no changes in psychiatric medications within the prior three months, and as confirmed by clinical interview during the screening phase. (Subjects who are currently hospitalized or have been hospitalized in the past three months for acute cocaine intoxication or withdrawal but who are otherwise psychiatrically stable as defined above are eligible for inclusion.)
* Females must be of non-child bearing potential or on appropriate contraceptive and not breast-feeding.
* Females must have a negative serum beta HCG at screening.
* The subject or his/her legal representative must provide informed, written consent.

Exclusion Criteria:

* Females who are pregnant or lactating
* Concurrent participation or participation within the prior 30 days in any study involving investigational medications
* Current diagnosis of Schizophrenia, Schizoaffective Disorder, or Bipolar Disorder
* Use of any antipsychotic medication within the prior three months
* History of idiopathic orthostatic hypotension, or sensitivity to the hypotensive effects of antipsychotic medication
* Angina pectoris or myocardial infarction in the 6 months prior to screening
* Persistent standing heart rate >120bpm or supine tachycardia (heart rate > 100 bpm)
* Sustained cardiac arrhythmia or history of clinically significant cardiac arrhythmia
* Cataracts (as per medical history or examination)
* Known personal history of seizure disorder
* Known history of seizure disorder in first-degree relatives
* History of significant head trauma, defined as head trauma resulting in loss of consciousness for more than five minutes and/or neurological or cognitive sequelae
* Use of potent cytochrome P450 inhibitors or inducers within 14 days before the baseline visit or during treatment, including but not limited to the agents identified in the study protocol
* Barbiturate use (as per self report or positive findings for barbiturates on the screening urine drug assay)
* Evidence of any clinically relevant disease (e.g., renal or hepatic impairment, significant coronary artery disease, cerebrovascular disease, hepatitis B or C, or cancer) or any clinical finding that in the opinion of the investigator could potentially be negatively affected by study participation or that could potentially affect study participation is criterion for exclusion from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
score on a self-report measure of cocaine use at 6 weeks | after 6 weeks treatment
score on a self-report measure of cocaine cravings at 6 wks | after 6 weeks treatment
results from urine drug screens across 6 weeks | weekly

SECONDARY OUTCOMES:
addiction severity | after 6 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andre Tapp, M.D., Principal Investigator — VA Puget Sound Health Care System, Tacoma and Seattle, WA and University of Washington, Department of Psychiatry and Behavioral Sciences, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System, American Lake Division, Tacoma, Washington, United States